CLINICAL TRIAL: NCT03842813
Title: Safety and Performance Assessment of Coronary Drug-Eluting Stent CRE8 : Post-market Observationnal Study
Brief Title: Safety and Performance Assessment of Drug-Eluting Stent CRE8 in Diabetic Patients
Acronym: EVALU8
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alvimedica Medical Technologies France (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02663-52
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Diabetes; Coronaropathy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: DES-CRE8 — Polymer-free Amphilimus™ (Sirolimus + Fatty Acid) eluting coronary stent. The absence of the polymer minimizes the risk of inflammation/thrombosis, while the propriety formulation enhances drug absorption.

SUMMARY:
The study is a 'real-world' study which evaluates the safety and performance of the coronary DES-CRE8 in diabetic patients.

As routine care, each patient will be followed until 12 months after stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old,
* patient informed and agreed to participate,
* patient with one or more lesions treated with one or more coronary stent CRE8,
* patient with a diabete insulin dependent or non-insulin dependant.

Exclusion Criteria:

* pregnant or breast-feading women,
* patient who refused to participate,
* patient with another lesion treated during the same intervention with a balloon alone or with another stent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation to the study will be proposed to all diabetic patients corresponding to the inclusion and exclusion criteria after implantation of one or more coronary stent CRE8.
  Patients will be consecutively included to limit selection bias.
Sampling Method: Probability Sample
Enrollment: 1030 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is Target Lesion Failure (TLF) rate at 1 year | 1 year post implantation
  The TLF is defined as cardiac deaths, heart attack in relation with the target vessel or revascularization of the target lesion.
  If a patient has at least one of these events, he will be considered as TLF.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) at 1 year | 1 year
  MACE are defined as: revascularization of the target lesion, heart attack or cardiac deaths.
Non cardiac deaths at 1 year | 1 year
  Non cardiac deaths at 1 year
Stent thrombosis at 1 year | 1 year
  Certain or probable stent thrombosis
Major Adverse Cardiac Events (MACE) at 1 year in the sub-group of patients with a short planned dual-therapy | 1 year
  MACE are defined as: revascularization of the target lesion, heart attack or cardiac deaths.
Non cardiac deaths at 1 year in the sub-group of patients with a short planned dual-therapy | 1 year
  Non cardiac deaths at 1 year
Stent thrombosis at 1 year in the sub-group of patients with a short planned dual-therapy | 1 year
  Certain or probable stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Julien Vandenwildenberg, Study Chair — Alvimedica Medical France
Locations (22):
- France (22):
  - Clinique de l'Europe, Amiens
  - Centre Hospitalier Avignon, Avignon
  - Centre Hospitalier Beauvais, Beauvais
  - Clinique Convert, Bourg-en-Bresse
  - Centre Hospitalier Brive, Brive-la-Gaillarde
  - Centre Hospitalier Chartres, Chartres
  - Hôpital Schweitzer, Colmar
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - Hôpital Privé de Bourgogne, Dijon
  - Hôpital Simone Veil, Eaubonne
  - Clinique Pasteur, Essey-lès-Nancy
  - Centre Hospitalier Gonesse, Gonesse
  - Centre Hospitalier Universitaire Grenoble, Grenoble
  - Centre Hospitalier Haguenau, Haguenau
  - Centre Hospitalier Saint-Joseph Saint-Luc, Lyon
  - Clinique Pont de Chaumes, Montauban
  - Centre Hospitalier Pau, Pau
  - Clinique Saint-Hilaire, Rouen
  - Centre Hospitalier Saint-Quentin, Saint-Quentin
  - Clinique Saint-Joseph, Trélazé
  - Centre Hospitalier Valence, Valence
  - Centre Hospitalier Vannes, Vannes

IPD SHARING:
Plan to Share IPD: No